CLINICAL TRIAL: NCT06106529
Title: A Randomized Intrapatient Cross-over Study to Assess the Efficacy of Oxybutynin Versus Venlafaxine in Reducing Hot Flashes in Women Using Endocrine Therapy After Breast Cancer.
Brief Title: REDucing Hot FLASHes in Women Using Endocrine Therapy.
Acronym: REDFLASH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Reinier de Graaf Groep (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REDFLASH2023-004
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Hot Flash Due to Medication
MeSH Terms: conditions — Breast Neoplasms | interventions — oxybutynin; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Venlafaxine (Experimental): In this open-label randomized controlled intrapatient cross-over study patients are randomly assigned to one of the two treatment groups.
  After a one week baseline period, group 1 starts with venlafaxine 37.5 mg once daily for 7 days followed by 75 mg once daily for 5 weeks followed by a two-week wash-out period (no medication), hereafter the group starts with oxybutynin 5 mg twice per day for 6 weeks total.
  Interventions: Drug: Oxybutynin; Drug: Venlafaxine
- Oxybutynin (Experimental): After a one week baseline period, group 2 starts with oxybutynin 5 mg twice per day for 6 weeks total followed by a two-week wash-out period (no medication), hereafter the group starts with venlafaxine 37.5 mg once daily for 7 days followed by 75mg once daily for 5 weeks.
  Interventions: Drug: Oxybutynin; Drug: Venlafaxine

INTERVENTIONS:
Drug: Oxybutynin — Oxybutynin 5 mg twice per day for 6 weeks
Drug: Venlafaxine — Venlafaxine 37.5 mg once daily for 7 days followed by 75 mg once daily for 5 weeks

SUMMARY:
The goal of this randomized intrapatient cross-over study is to assess the efficacy of oxybutynin versus venlafaxine in reducing hot flashes in women using endocrine therapy after breast cancer.

The objectives it aims to answer are:

* To assess the efficacy of oxybutynin versus venlafaxine in reducing hot flashes in women using endocrine therapy after breast cancer
* To assess side effects of oxybutynin versus venlafaxine.
* To assess the personal preference of women for oxybutynin versus venlafaxine in reducing hot flashes.
* To assess quality of life of women when reducing hot flashes in women using endocrine therapy after breast cancer.

Participants will fill-out a patient diary during 15 weeks total on a daily basis and receive an (online) questionnaire three times total.

Researchers will compare two groups (venlafaxine group versus oxubutynine group) to assess its efficacy concerning hot flashes.

ELIGIBILITY:
Inclusion Criteria:

* Pre-, peri- or postmenopausal women of 18 years or above;
* Indication for endocrine therapy and already started with tamoxifen, aromatase inhibitors or luteinizing hormone-releasing hormone analogues for at least 4 weeks and planning to continue for the duration of the study;
* Experiencing hot flashes with a minimum of 14 per week for at least 1 month and desire to start a pharmacologic intervention.

Exclusion Criteria:

* Pregnant;
* Breast feeding;
* Patients who receive chemotherapy or immunotherapy/HER2 antibodies within the prior 8 weeks, and patients scheduled for chemotherapy during the study period;
* Palliative setting;
* Use of venlafaxine or any other antidepressants, also including St. John's wort within the previous year;
* Creatinine clearance < 30 ml/min;
* Liver cirrhosis;
* Use of gabapentin and/or calcium channel antagonists within 2 weeks of study entry;
* Use of oxybutynin before study entry;
* Use of any other substances or therapies for the treatment of hot flashes, for instance acupuncture.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number and severity of hot flashes | 15 weeks total
  Number and severity of hot flashes during 6-weeks of therapy measured by the Hot Flash Diary.

SECONDARY OUTCOMES:
Quality of life and health status | 15 weeks total
  Quality of life and health status at baseline and after 6 weeks of treatment measured by the EORTC-QLQ-C30
Adverse effects of treatments | 15 weeks total
  Adverse effects of treatments weekly measured by the National Cancer Institute Common Toxicity Criteria scale, version 5
Sleep quality | 15 weeks total
  Sleep quality at baseline and after 6 weeks of treatment measured by the Groningen Sleep Quality Scale (GSQ)
Anxiety and depression | 15 weeks total
  Anxiety and depression measured at baseline and after 6 weeks of treatment with the Hospital Anxiety and Depression Scale (HADS)
Sexual function | 15 weeks total
  Sexual function measured at baseline and after 6 weeks of treatment with the Sexual Activity Questionnaire (SAQ)
Cognitive function | 15 weeks total
  Cognitive function measured at baseline and after 6 weeks of treatment with the 6-item cognitive impairment test (6-CIT)
Adherence | 15 weeks total
  Ask patients the following question after 6 weeks of treatment: 'Would you like to continue the endocrine therapy for the recommended duration of therapy taking the current medication (oxybutynin or venlafaxine) given the number and severity of hot flashes you experience during the last week?'
Preference | 15 weeks total
  Ask patients the following question after 6 weeks of the final treatment: 'Do you have a preference taking the medication from study period 1 or study period 2?'

CONTACTS AND LOCATIONS:
Overall Officials: Lemonitsa Mammatas, PhD, Principal Investigator — Reinier De Graaf Ziekenhuis
Locations (1):
- Reinier de Graaf Gasthuis, Delft, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, anonymised database and study results may be available on request, after assessment of the reason for request by the study investigators.
Supporting Information: Study Protocol, SAP, CSR